CLINICAL TRIAL: NCT01511887
Title: Evaluation of the Safety and Efficacy of Oral Ibuprofen in Term 20-28 Days Old Newborns Referred to Bandar Abbass Children Hospital in 2011
Brief Title: Safety and Efficacy of Ibuprofen in Term Newborns With Patent Ductus Arteriosus (PDA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hamidreza Mahboobi, Principal Investigator, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ibuprofen in PDA
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent Ductus Arteriosus; PDA; Term newborns; Ibuprofen
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Ibuprofen (Experimental): 10mg/kg oral ibuprofen followed by two 5mg/kg in 12 hours intervals. If there was no improvement after first cycle of treatment this treatment was repeated.
  Interventions: Drug: Oral Ibuprofen
- No treatment (No Intervention): No treatment

INTERVENTIONS:
Drug: Oral Ibuprofen — 10mg/kg oral ibuprofen followed by two 5mg/kg in 12 hours intervals. If there was no improvement after first cycle of treatment this treatment was repeated.
  Other Names: Advil
  Arms: Oral Ibuprofen

SUMMARY:
The aim of current study is to evaluate the efficacy and safety of oral Ibuprofen in term 20-28 days old newborn referred to Bandarabbas children' hospital in 2011.

DETAILED DESCRIPTION:
Patent Ductus Arteriosus (PDA) accounts for about 10% of Congenital Heart Disease. Surgical treatment in PDA is associated with higher rate of complication than pharmacologic treatment. Efficacy of Ibuprofen is shown in preterm and low birth weights newborn with PDA. Studies in term neonates after the first days of birth are rare. The aim of current study is to evaluate the efficacy and safety of oral Ibuprofen in term 20-28 days old newborn referred to Bandarabbas children' hospital in 2011.

ELIGIBILITY:
Inclusion Criteria:

* Term newborn (37 weeks of gestation or more)
* Age between 20-28 days
* confirmed diagnosis of PDA by echocardiography by pediatric cardiologist

Exclusion Criteria:

* Asphyxia
* Hemorrhage
* Platelet count < 150000
* renal or gastrointestinal malformations
* associated congenital heart disease

Ages: 20 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
PDA closure after 1 week | 1 weeks after treatment
  PDA closure after 1 week of treatment based on echocardiography
PDA closure after two weeks | 2 weeks after treatment
  PDA closure two weeks after treatment based on echocardiography

SECONDARY OUTCOMES:
Drug side effects | two weeks after treatment
  hemorrhage, abdominal distention, oliguria

CONTACTS AND LOCATIONS:
Overall Officials: Hamidreza Mahboobi, MD, Principal Investigator — Hormozgan University of Medical Sciences (HUMS)
Locations (1):
- Hormozgan University of Medical Sciences, Bandar Abbas, Hormozgan, Iran